CLINICAL TRIAL: NCT01589991
Title: Anticaries Potential and Fluorosis Risk From Different Fluoride Toothpastes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Livia Maria Andaló Tenuta, Assistant Professor, Biochemistry and Cariology, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FOPBioq002
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Dental Caries; Dental Fluorosis
Keywords: toothpastes; bioavailability; sodium fluoride; monofluorphosphate; low-fluoride
MeSH Terms: conditions — Dental Caries; Fluorosis, Dental | interventions — Toothpastes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Non-fluoride toothpaste (Placebo Comparator)
  Interventions: Drug: Toothpaste
- Toothpaste 550 µg F/g (NaF/SiO2) (Experimental)
  Interventions: Drug: Toothpaste
- Toothpaste 1100 µg F/g (NaF/SiO2) (Experimental)
  Interventions: Drug: Toothpaste
- Toothpaste 1450 µg F/g (MFP/CaCO3) (Experimental)
  Interventions: Drug: Toothpaste

INTERVENTIONS:
Drug: Toothpaste — The volunteers brushed their teeth with 0.3 g of the assigned toothpastes, 3x/day.

SUMMARY:
Fluoride toothpaste has been associated not only with declining dental caries prevalence but also with an increase in dental fluorosis. In the balance of benefits/risks of fluoride toothpaste use, the purpose of this study is to evaluate the availability of fluoride concentration in the mouth (biofilm fuild), as an indicator of fluoride benefits (anticaries effect), and the fluoride concentration in urine, as an indicator of fluoride absorption from ingested toothpastes (with potential to cause dental fluorosis), in a sample of young Brazilian children using toothpaste formulations representative of those available and most used by this age-group.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Good oral health

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Fluoride concentration in biofilm fluid | 30min
  Remants of dental plaque (biofilm) will be collected 30 min after brushing with the toothpastes, the fluid will be separated from the solids by centrifugation and the fluoride concentration in the biofilm fluid will be determined by a fluoride electrode adapted for microanalysis.
Urinary fluoride excretion | 8h
  Urine will be collected at two time-points, either before the use of the toothpaste or at the last day of use, in each experimental phase. Fluoride concentration was determined by an inverted ion-specific fluoride electrode and fluoride excretion will be measured by fluoride/cratinine ratio (mg F/mg creatinine).

SECONDARY OUTCOMES:
Fluoride concentration in biofilm solid | 30min
  Remants of dental plaque (biofilm) will be collected 30 min after brushing with the toothpastes, the fluid will be separated from the solids by centrifugation and the fluoride concentration in the biofilm solids will be determined after acid extraction using a fluoride electrode adapted for microanalysis.
Fluoride concentration in saliva | 30min
  Non-stimulated saliva will be collected at 0 (immediately before toothbrushing), 7, 15 and 30 min after toothbrushing. Fluoride concentration in saliva will be determined by a ion-specific fluoride electrode, adapted for microanalysis.
Amount of toothpaste ingested | January 2013 to July 2013
  Determination of amount of toothpaste ingested after one simulated brushing.

CONTACTS AND LOCATIONS:
Overall Officials: Livia MA Tenuta, PhD, Study Chair — Piracicaba Dental School, University of Campinas
Locations (1):
- Piracicaba Dental School, University of Campinas, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Background] Cury JA, do Amaral RC, Tenuta LM, Del Bel Cury AA, Tabchoury CP. Low-fluoride toothpaste and deciduous enamel demineralization under biofilm accumulation and sucrose exposure. Eur J Oral Sci. 2010 Aug;118(4):370-5. doi: 10.1111/j.1600-0722.2010.00745.x. PMID 20662910
- [Background] Lima TJ, Ribeiro CC, Tenuta LM, Cury JA. Low-fluoride dentifrice and caries lesion control in children with different caries experience: a randomized clinical trial. Caries Res. 2008;42(1):46-50. doi: 10.1159/000111749. Epub 2007 Nov 27. PMID 18042987
- [Background] Cury JA, Tenuta LM, Ribeiro CC, Paes Leme AF. The importance of fluoride dentifrices to the current dental caries prevalence in Brazil. Braz Dent J. 2004;15(3):167-74. doi: 10.1590/s0103-64402004000300001. Epub 2005 Mar 18. PMID 15798817
- [Background] Paes Leme AF, Dalcico R, Tabchoury CP, Del Bel Cury AA, Rosalen PL, Cury JA. In situ effect of frequent sucrose exposure on enamel demineralization and on plaque composition after APF application and F dentifrice use. J Dent Res. 2004 Jan;83(1):71-5. doi: 10.1177/154405910408300114. PMID 14691117
- [Background] Cury JA, Francisco SB, Simoes GS, Del Bel Cury AA, Tabchoury CP. Effect of a calcium carbonate-based dentifrice on enamel demineralization in situ. Caries Res. 2003 May-Jun;37(3):194-9. doi: 10.1159/000070444. PMID 12740543
- [Background] Cury JA, Simoes GS, Del Bel Cury AA, Goncalves NC, Tabchoury CP. Effect of a calcium carbonate-based dentifrice on in situ enamel remineralization. Caries Res. 2005 May-Jun;39(3):255-7. doi: 10.1159/000084807. PMID 15914990
- [Background] Cury JA, Oliveira MJ, Martins CC, Tenuta LM, Paiva SM. Available fluoride in toothpastes used by Brazilian children. Braz Dent J. 2010;21(5):396-400. doi: 10.1590/s0103-64402010000500003. PMID 21180793
- [Background] Martins CC, Oliveira MJ, Pordeus IA, Cury JA, Paiva SM. Association between socioeconomic factors and the choice of dentifrice and fluoride intake by children. Int J Environ Res Public Health. 2011 Nov;8(11):4284-99. doi: 10.3390/ijerph8114284. Epub 2011 Nov 10. PMID 22163207